CLINICAL TRIAL: NCT05892796
Title: Prediction of Morbidity and Mortality With Medical Pre-Operative Fitness Assessment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasmeen Abdelshafy Ebrahim, Investigator, Assiut University
Other Study IDs: mPOFA
Record Dates: First submitted 2023-05-16; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Perioperative Medical Fitness Assessment
Keywords: Fitness Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim to measure the predictability of medical pre -Operative Fitness Assessment to the actual rates of morbidity and mortality related to surgery in Assiut university Hospital.

DETAILED DESCRIPTION:
Perioperative morbidity and mortality remain the mostly important barrier to surgical interventions worldwide. Therefor, decision making relies upon accurate risk Assessment to be balanced with hoped benefit.

For elective surgeries, multiple clinical tools have been used to Assessment perioperative Fitness, but with limited applicability. For instance, the american society of anesthesiologists phesical status score (ASA-PS) does not consider the type of surgery, nor the patient's age.

The physiological and Operative severity score for the enumeration of mortality (POSSUM) evaluates the intra-operative difficulties, limiting the preoperative prediction.

Recently, researchers layer and his colleagues at University Hospital Bonn, modified the preoperative score to Predict Postoperative Mortality (POSPOM) to be applied in daily practice.

In investigator 's practice, Assiut university Hospitals already have a Pre-Operative Fitness Assessment (POFA) clinical and investigator aim to adapt and evaluate the POSPOM system in investigator' s practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years old ) preparing for elective intervention.

Exclusion Criteria:

* those who do not require anaesthesia Those who did not undergo surgery

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults >18 Inclusion Criteria:
  * Adults (>18 years old ) preparing for elective intervention
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidance of 22 adverse events according to the Eurepian perioperative clinical outcom definitions | Baseline
  Follow up of preoperative medically diseased patients after surgery to detect outcoms

REFERENCES:
- [Background] Conrad C, Eltzschig HK. Disease Mechanisms of Perioperative Organ Injury. Anesth Analg. 2020 Dec;131(6):1730-1750. doi: 10.1213/ANE.0000000000005191. PMID 33186161
- [Background] Eyob B, Boeck MA, FaSiOen P, Cawich S, Kluger MD. Ensuring safe surgical care across resource settings via surgical outcomes data & quality improvement initiatives. Int J Surg. 2019 Dec;72S:27-32. doi: 10.1016/j.ijsu.2019.07.036. Epub 2019 Aug 5. PMID 31394278
- [Background] Sankar A, Johnson SR, Beattie WS, Tait G, Wijeysundera DN. Reliability of the American Society of Anesthesiologists physical status scale in clinical practice. Br J Anaesth. 2014 Sep;113(3):424-32. doi: 10.1093/bja/aeu100. Epub 2014 Apr 11. PMID 24727705
- [Background] Copeland GP, Jones D, Walters M. POSSUM: a scoring system for surgical audit. Br J Surg. 1991 Mar;78(3):355-60. doi: 10.1002/bjs.1800780327. PMID 2021856
- [Background] Le Manach Y, Collins G, Rodseth R, Le Bihan-Benjamin C, Biccard B, Riou B, Devereaux PJ, Landais P. Preoperative Score to Predict Postoperative Mortality (POSPOM): Derivation and Validation. Anesthesiology. 2016 Mar;124(3):570-9. doi: 10.1097/ALN.0000000000000972. PMID 26655494
- [Background] Layer YC, Menzenbach J, Layer YL, Mayr A, Hilbert T, Velten M, Hoeft A, Wittmann M. Validation of the Preoperative Score to Predict Postoperative Mortality (POSPOM) in Germany. PLoS One. 2021 Jan 27;16(1):e0245841. doi: 10.1371/journal.pone.0245841. eCollection 2021. PMID 33503043